CLINICAL TRIAL: NCT04807010
Title: PROARTE -PROstate ARTery to Reduce the Symptoms of Benign Prostatic Hyperplasia
Acronym: PROARTE
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Society of Interventional Radiology Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2021-03-11; First posted 2021-03-19 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Benign Prostatic Hyperplasia; Lower Urinary Tract Symptoms
Keywords: Prostate artery embolization; Benign Prostatic Hyperplasia; Lower Urinary Tract Symptoms; Quality of Life
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients and those recording response will be blinded to cohort allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prostate artery embolization (Active Comparator)
  Interventions: Procedure: Prostate Artery Embolization
- Sham (Sham Comparator)
  Interventions: Procedure: Prostate Artery Embolization; Procedure: Sham Prostate Artery Embolization

INTERVENTIONS:
Procedure: Prostate Artery Embolization — Prostate artery embolization reduces symptoms from benign prostatic hyperplasia by delivering embolic materials to the prostate through the prostatic arteries.
Procedure: Sham Prostate Artery Embolization — Angiogram without embolization initially. At 6 months patients will be allowed to crossover to prostate artery embolization.
  Arms: Sham

SUMMARY:
This is a trial to demonstrate the superiority of prostate artery embolization (PAE) over sham procedure in men with benign prostatic hyperplasia (BPH) induced lower urinary tract symptoms (LUTS). The trial will aim to enroll 108 patients at a 2:1 allocation over a 2 year period.

ELIGIBILITY:
Inclusion Criteria:

* • Men ≥45 and ≤90 years presenting with benign prostatic hyperplasia with symptoms for at least 6 months that are refractory to medical management or in whom medications are contraindicated, not tolerated, or refused.

  * International Prostate Symptom Score (I-PSS) score 14 or greater.
  * Quality of Life (QoL) score ≥ 3
  * Peak urinary flow (Qmax) less than or equal to 12 mL/s with void volume >125mL.
  * Prostate volume greater than 30 cc as determined by ultrasound, MRI, or CT.
  * Personal risk <40% based on the University of Texas San Antonio prostate cancer risk calculator or having a negative prostate biopsy for cancer within the last 24 months.
  * Able to provide written consent.
  * Not participating in any other investigational drug or device studies.

Exclusion Criteria:

* • History of biopsy-proven prostate cancer

  * Renal insufficiency (glomerular filtration rates (GFR) less than 40mL/min/1.73 m2 who are not already on dialysis)
  * Prior prostate surgery or intervention, including trans-urethral resection of the prostate, balloon dilation, stent implantation, laser prostatectomy, radiation, UroLift®, or hyperthermia
  * Other bladder or urethral pathology requiring therapy, either in the past or currently, including neurogenic bladder, sphincteric abnormalities, bladder cancer, or other causes of bladder atonia.
  * Other causes of urinary obstruction, such as strictures of urethra or ureters, not related to BPH
  * Current decompensated congestive heart failure, uncontrolled diabetes mellitus, significant respiratory disease, or known immunosuppression.
  * Neurological disease, including multiple sclerosis, amyotrophic lateral sclerosis, Parkinson's disease, and previous spinal nerve surgery
  * Patients with platelet count <50,000/μL or International Normalized Ratio (INR) >1.8, unless corrected for the procedure
  * Active urinary tract infection. Patients must have a negative culture within 7 days of the procedure.
  * Allergy to iodinated contrast agents unless pre-treated by corticosteroids.
  * Acute urinary retention.
  * Post void residual (PVR) > 250 mL with urodynamic evidence of atonic bladder. Patients with a PVR >250 but urodynamic testing consistent with obstruction will be allowed.
  * Bladder stone within three months prior to the procedure.
  * Hematuria not evaluated by Urologist for causes other than BPH.
  * Previous rectal surgery (excluding hemorrhoidectomy) or history of rectal disease.
  * Prior pelvic irradiation or radical pelvic surgery.

Imaging exclusion criteria:

• Internal iliac artery occlusion as determined by either CT or MRI.

Ages: 45 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients must be male, as they are the only ones who suffer from BPH induced LUTS
Enrollment: 108 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
International Prostate Symptom Score | 6 months
  A survey accessing patient symptomology from BPH induced LUTS

SECONDARY OUTCOMES:
International Prostate Symptom Score | 1, 3, 6, 9, 12, 24, 36 months
  A survey accessing patient symptomology from BPH induced LUTS
Quality of Life | 1, 3, 6, 9, 12, 24, 36 months
  A survey accessing quality of life impact on patients from BPH induced LUTS.
Maximal urinary flow rate change from baseline | 6, 12, 24, and 36 months
  Maximal flow rate of urine stream
Post void residual change from baseline | 6, 12, 24, and 36 months
  Post void residual measures the volume of urine remaining in the bladder after complete emptying.
International Index of Erectile Function questionnaire (IIEF) | 1, 3, 6, 9, 12, 24, 36 months
  A questionnaire designed to asses erectile function
Freedom from secondary intervention to treat BPH | 1, 3, 6, 9, 12, 24, 36 months
  Recording of other surgical/procedural treatments with each procedure being recorded as an event.
Ejaculatory function | 3, 6, 9, 12, 24, 36 months
  Ejaculatory function will be assessed utilizing a four item questionnaire.
Urinary Continence | 1, 6, and 12 months
  Urinary Continence will be assessed using a 2 item questionnaire
Number of hospital days | 1 month
  Number of hospital days following the procedure will be recorded
Recover experience | 1 month
  Recover experience will be assessed using a quality of recovery visual analog scale
Adverse events | 7 days and 1, 3, 6, 9, 12, 24, 36 months
  All procedure related adverse events will be recoreded

CONTACTS AND LOCATIONS:
Overall Officials: Shamar Young, MD, Principal Investigator — University of Minnesota; Jafar Golzarian, MD, Principal Investigator — University of Minnesota

IPD SHARING:
Plan to Share IPD: Undecided